CLINICAL TRIAL: NCT06058377
Title: Phase III Trial Of Neoadjuvant Durvalumab (NSC 778709) Plus Chemotherapy Versus Chemotherapy Alone For Adults With MammaPrint High 2 Risk (MP2) Hormone Receptor (HR) Positive / Human Epidermal Growth Factor Receptor (HER2) Negative Stage II-III Breast Cancer
Brief Title: Adding an Immunotherapy Drug, MEDI4736 (Durvalumab), to the Usual Chemotherapy Treatment (Paclitaxel, Cyclophosphamide, and Doxorubicin) for Stage II-III Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-04566; NCI-2023-04566 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2206 (Other: SWOG); S2206 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-09-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; HER2-Negative Breast Carcinoma; Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: interventions — Specimen Handling; Cyclophosphamide; Doxorubicin; durvalumab; Immunoglobulin G; Disulfides; Genetic Testing; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Step 1 (MammaPrint testing) (Experimental): Patients without a known MP2 score undergo MammaPrint testing on a previously-collected tissue sample. Patients with MP2 score proceed to STEP 2
  Interventions: Other: Genetic Testing
- Step 2, Arm 1 (chemotherapy) (Active Comparator): Patients receive paclitaxel IV on days 1 and 8 of each cycle. Treatment repeats every 14 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive doxorubicin IV and cyclophosphamide IV on day 1 of each cycle. Treatment repeats every 14 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo mammography during screening (STEP 1). Patients have the option to also undergo collection of tumor tissue during initial biopsy (STEP 1) and at SOC surgery and undergo collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cyclophosphamide; Drug: Doxorubicin; Procedure: Mammography; Drug: Paclitaxel; Other: Quality-of-Life Assessment
- Step 2, Arm 2 (chemotherapy, durvalumab) (Experimental): Patients receive paclitaxel IV on days 1 and 8 of each cycle and durvalumab IV over 60 minutes on day 1 of cycles 1, 3, and 5. Treatment repeats every 14 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive doxorubicin IV and cyclophosphamide IV on day 1 of each cycle, and durvalumab IV over 60 minutes on day 1 of cycles 7 and 9. Treatment repeats every 14 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo mammography during screening (STEP 1). Patients have the option to also undergo collection of tumor tissue during initial biopsy (STEP 1) and at SOC surgery and undergo collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Durvalumab; Procedure: Mammography; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo optional collection of tissue and/or blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Step 2, Arm 1 (chemotherapy); Step 2, Arm 2 (chemotherapy, durvalumab)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Step 2, Arm 1 (chemotherapy); Step 2, Arm 2 (chemotherapy, durvalumab)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Step 2, Arm 1 (chemotherapy); Step 2, Arm 2 (chemotherapy, durvalumab)
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Step 2, Arm 2 (chemotherapy, durvalumab)
Other: Genetic Testing — Undergo MammaPrint testing
  Other Names: Genetic Analysis; Genetic Examination; Genetic Test
  Arms: Step 1 (MammaPrint testing)
Procedure: Mammography — Undergo mammography
  Other Names: MG
  Arms: Step 2, Arm 1 (chemotherapy); Step 2, Arm 2 (chemotherapy, durvalumab)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Step 2, Arm 1 (chemotherapy); Step 2, Arm 2 (chemotherapy, durvalumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Step 2, Arm 1 (chemotherapy); Step 2, Arm 2 (chemotherapy, durvalumab)

SUMMARY:
This phase III trial compares the addition of an immunotherapy drug (durvalumab) to usual chemotherapy versus usual chemotherapy alone in treating patients with MammaPrint High 2 Risk (MP2) stage II-III hormone receptor positive, HER2 negative breast cancer. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as paclitaxel, doxorubicin, and cyclophosphamide work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. There is some evidence from previous clinical trials that people who have a MammaPrint High 2 Risk result may be more likely to respond to chemotherapy and immunotherapy. Adding durvalumab to usual chemotherapy may be able to prevent the cancer from returning for patients with MP2 stage II-III hormone receptor positive, HER2 negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare breast cancer event-free survival between participants randomized to standard of care neoadjuvant chemotherapy alone versus standard of care neoadjuvant chemotherapy concurrent with durvalumab.

SECONDARY OBJECTIVES:

I. To compare pathologic complete response rates (ypT0/is, ypN0) in participants randomized to standard of care chemotherapy alone versus (vs.) standard of care neoadjuvant chemotherapy concurrent with durvalumab.

II. To compare residual cancer burden distribution between participants randomized to standard of care neoadjuvant chemotherapy vs. standard of care neoadjuvant chemotherapy concurrent with durvalumab.

III. To compare distant relapse-free survival between participants randomized to standard of care neoadjuvant chemotherapy vs. standard of care neoadjuvant chemotherapy concurrent with durvalumab.

IV. To compare overall survival between participants randomized to standard of care neoadjuvant chemotherapy vs. standard of care neoadjuvant chemotherapy concurrent with durvalumab.

V. To compare the frequency and severity of toxicities between participants randomized to standard of care neoadjuvant chemotherapy vs. standard of care neoadjuvant chemotherapy concurrent with durvalumab among those who initiate the assigned treatment.

PRIMARY QUALITY OF LIFE (QOL) OBJECTIVES:

I. To compare the change in fatigue (Patient Reported Outcomes Measurement Information System [PROMIS] Fatigue) experienced by participants randomized to neoadjuvant durvalumab plus chemotherapy vs. participants randomized to chemotherapy alone at completion of active treatment (at 20 weeks from baseline).

II. To compare the change in global physical health (PROMIS Global Health) experienced by participants randomized to neoadjuvant durvalumab plus chemotherapy vs participants randomized to chemotherapy alone at completion of active treatment (at 20 weeks from baseline).

SECONDARY QOL OBJECTIVES:

I. To compare the change in fatigue and global physical health experienced by participants randomized to neoadjuvant durvalumab plus chemotherapy vs participants randomized to chemotherapy alone during treatment (at 12 weeks from baseline).

II. To compare the changes in global physical health and fatigue subsequent to treatment (at years 1 and 2) between the two randomized study arms.

III. To compare the changes in global mental health (PROMIS Global Health) during active treatment (weeks 12, 20) and subsequent to treatment (at years 1 and 2) between the two randomized study arms.

IV. To compare the severity and frequency of treatment-related symptoms using Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) items (diarrhea, nausea, cough, shortness of breath, rash, and musculoskeletal pain) over time experienced by participants receiving neoadjuvant durvalumab plus chemotherapy versus chemotherapy alone.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

STEP 1: Patients without a known MP2 score undergo MammaPrint testing on a previously-collected tissue sample. Patients with MP2 score proceed to STEP 2.

STEP 2: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive paclitaxel intravenously (IV) on days 1 and 8 of each cycle. Treatment repeats every 14 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive doxorubicin IV and cyclophosphamide IV on day 1 of each cycle. Treatment repeats every 14 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive paclitaxel IV on days 1 and 8 of each cycle and durvalumab IV over 60 minutes on day 1 of cycles 1, 3, and 5. Treatment repeats every 14 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive doxorubicin IV and cyclophosphamide IV on day 1 of each cycle, and durvalumab IV over 60 minutes on day 1 of cycles 7 and 9. Treatment repeats every 14 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

All patients also undergo mammography during screening (STEP 1). Patients have the option to also undergo collection of tumor tissue during initial biopsy (STEP 1) and at standard of care (SOC) surgery and undergo collection of blood samples throughout the study.

After completion of study treatment, patients are followed until death or 10 years, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1: REGISTRATION (SCREENING): Participants must have histologically confirmed estrogen receptor (ER) positive and/or progesterone receptor (PR) positive (hormone receptor positive) and HER2 negative breast cancer, as per American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines

  * NOTE: Participants with HER2 positive disease by ASCO CAP guidelines are ineligible. HER2 negative and HER2 low or equivocal cases as per ASCO CAP guidelines that do not receive HER2 targeted therapy are eligible
* STEP 1: REGISTRATION (SCREENING): Participants must have clinical stage II or III breast cancer

  * NOTE: Participants with inflammatory breast cancer are eligible
  * NOTE: Participants with occult (i.e. undetectable) primary breast cancer with axillary nodal involvement are not eligible, as MammaPrint testing has not been validated on tissue obtained from an axillary lymph node
* STEP 1: REGISTRATION (SCREENING): Participants must not have metastatic disease (i.e., must be clinically M0 or Mx) Systemic staging studies with imaging should follow routine practice as per National Comprehensive Cancer Network (NCCN) and ASCO guidelines
* STEP 1: REGISTRATION (SCREENING): Participants must not have locally recurrent breast cancer
* STEP 1: REGISTRATION (SCREENING): Participants with multifocal disease in the same breast or synchronous bilateral primary tumors are eligible, however, all tumors that are biopsied must be hormone receptor positive and HER2 negative per ASCO CAP guidelines and at least one of the tumors must be MammaPrint High-2. MammaPrint can be performed sequentially on biopsies as it is sufficient to have MammaPrint High 2 status on at least one of the lesions

  * NOTE: Biopsy of multiple lesions in the same breast is not required if the clinical presentation is consistent with a single disease process that is multifocal in nature. However, if there is clinical suspicion of two distinct primary breast malignancies, additional biopsies should be pursued
* STEP 1: REGISTRATION (SCREENING): Participants must have either adequate tissue available to submit on-study or a prior known MammaPrint Index Score that is MP2 status

  * Submitting tissue for on-study MammaPrint testing:

    * Participants must have a minimum of ten, unstained formalin-fixed paraffin-embedded (FFPE) slides (4-5 micron thickness) available from initial tumor biopsy for MammaPrint assessment

      * NOTE: Participants must agree to have this tissue submitted to Agendia for MammaPrint Index Scoring and to have subsequent results disclosed to Southwest Oncology Group (SWOG) Cancer Research Network OR
  * Submitting prior known MammaPrint Index Score:

    * If a MammaPrint Index Score report from within the last 12 weeks is already known and is MP2 status, the participant must be registered to Step 2 immediately following Step 1 registration provided they meet all other criteria. MP2 status is defined as a MammaPrint Index score between negative 1.0 and negative 0.57 (-1.0 to -0.57, including negative 1.0 and negative 0.57) tested from initial tumor biopsy

      * NOTE: Participants must agree to have their commercial MammaPrint Index Score disclosed to SWOG Cancer Research Network
      * NOTE: Participants with prior known MammaPrint result that is not MP2 status should not be enrolled to either step of this study
      * NOTE: Participants enrolling with known MP2 status (i.e. MP already obtained as routine care) must only sign the treatment informed consent form. Screening consent is not required when MP2 status is known prior to study enrollment
* STEP 1: REGISTRATION (SCREENING): Participants must not have received any prior treatment for their current breast cancer, including chemotherapy, immunotherapy, biologic or hormonal therapy, and must be candidates for doxorubicin, paclitaxel, and durvalumab therapy
* STEP 1: REGISTRATION (SCREENING): Participants must be >= 18 years old at the time of registration
* STEP 1: REGISTRATION (SCREENING): Participants must have body weight > 30 kg
* STEP 1: REGISTRATION (SCREENING): Participants must have Zubrod Performance Status of 0-2
* STEP 1: REGISTRATION (SCREENING): Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* STEP 1: REGISTRATION (SCREENING): Participant must not have medical contraindications to receiving immunotherapy, including history of non-infectious pneumonitis that required steroids or active autoimmune disease that has required systemic treatment with disease modifying agents, corticosteroids or immunosuppressive drugs in the past two years. Replacement therapy (e.g. thyroxine for pre-existing hypothyroidism, insulin for type I diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Intra-articular steroid injections are allowed
* STEP 1: REGISTRATION (SCREENING): NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
  * For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
* STEP 2: RANDOMIZATION: Participants must have met all eligibility criteria for Step 1 Registration
* STEP 2: RANDOMIZATION: Participants must have MammaPrint High Risk 2 result

  * For participants submitting tissue for on-study MammaPrint testing:

    * Participants must be registered to Step 2: Randomization within 84 calendar days (12 weeks) after receiving an MP2 status from the MammaPrint Index score. MP2 status is defined as a MammaPrint Index score between negative 1.0 and negative 0.57 (-1.0 to -0.57, including negative 1.0 and negative 0.57) from initial tumor biopsy OR
  * Submitting commercial MammaPrint Index Score:

    * If a MammaPrint Index Score report from within the last 12 weeks is already known and is MP2 status, the participant must be registered to Step 2 immediately following Step 1 registration provided they meet all other criteria. MP2 status is defined as a MammaPrint Index score between negative 1.0 and negative 0.57 (-1.0 to -0.57, including negative 1.0 and negative 0.57) tested from initial tumor biopsy

      * NOTE: Participants without a MammaPrint High-Risk 2 score must not be registered to Step 2 Randomization
* STEP 2: RANDOMIZATION: Participants must not have received live vaccines within 28 days prior to study Step 2: Randomization. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Seasonal influenza vaccines and coronavirus disease 2019 (COVID-19) vaccines are allowed; however, intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated vaccines, and are not allowed
* STEP 2: RANDOMIZATION: Participants must not be planning to receive any concurrent non-protocol directed chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study
* STEP 2: RANDOMIZATION: Participant must have Zubrod Performance Status of 0-2
* STEP 2: RANDOMIZATION: Participants must not have a history of (non-infectious) pneumonitis that required steroids or evidence of active pneumonitis within two years prior to Step 2: Randomization
* STEP 2: RANDOMIZATION: Participants must not have active autoimmune disease that has required systemic treatment in the past two years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) prior to Step 2: Randomization. Replacement therapy (e.g. thyroxine for pre-existing hypothyroidism, insulin for type I diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Intra-articular steroid injections are allowed
* STEP 2: RANDOMIZATION: Participant must have a complete medical history and physical exam within 28 days prior to Step 2: Randomization
* STEP 2: RANDOMIZATION: Leukocytes >= 3 x 10^3/uL (within 28 days prior to Step 2: Randomization)
* STEP 2: RANDOMIZATION: Absolute neutrophil count >= 1.5 x 10^3/uL (within 28 days prior to Step 2: Randomization)
* STEP 2: RANDOMIZATION: Platelets >= 100 x 10^3/uL (within 28 days prior to Step 2: Randomization)
* STEP 2: RANDOMIZATION: Total bilirubin =< institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to Step 2: Randomization)
* STEP 2: RANDOMIZATION: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 × institutional ULN (within 28 days prior to Step 2: Randomization)
* STEP 2: RANDOMIZATION: Participants must have a calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to Step 2: Randomization
* STEP 2: RANDOMIZATION: Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* STEP 2: RANDOMIZATION: Participants must not have uncontrolled diabetes defined as hemoglobin A1c of 9.0% or greater, within 28 days prior to Step 2: Randomization
* STEP 2: RANDOMIZATION: Participants with history of human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have an undetectable viral load on the most recent test results obtained within 6 months prior to Step 2: Randomization
* STEP 2: RANDOMIZATION: Participants with history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on the most recent test results obtained while on suppressive therapy within 6 months prior to Step 2: Randomization, if indicated
* STEP 2: RANDOMIZATION: Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load on the most recent test results obtained within 6 months prior to Step 2: Randomization, if indicated
* STEP 2: RANDOMIZATION: Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method during protocol therapy and for 6 months following completion of protocol therapy with details provided as a part of the consent process and must have a negative pregnancy test at screening. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen. Participants should not breastfeed during protocol therapy and for 6 months following completion of protocol therapy
* STEP 2: RANDOMIZATION: Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the SWOG Specimen Tracking System
* STEP 2: RANDOMIZATION: Participants who can complete questionnaires in English, or Spanish must be offered the opportunity to participate in the Quality of Life study
* STEP 2: RANDOMIZATION: NOTE: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2: RANDOMIZATION: Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3680 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Breast cancer event-free survival (BC-EFS) | Up to 10 years after completion of study treatment
  Defined as the earliest occurrence of any of the following events: Local-regional or distant progression during neoadjuvant therapy or local/regional, or distant invasive breast tumor recurrence post-surgery, invasive ipsilateral breast tumor recurrence, new invasive contralateral breast cancer, or death from any cause. The primary analysis of BC-EFS is a log-rank test between the treatment arms with stratification by the three stratification factors. Additionally, Cox regression will be used to estimate the treatment hazard ratio and 95% confidence interval including the three stratification variables as terms in the model. Kaplan-Meier graphs will show BC-EFS descriptively over time and provide 5-year estimates and 95% confidence intervals. A forest plot will show whether the treatment effect varies over the stratification variables and other selected factors.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) rates | Up to 10 years after completion of study treatment
  Defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast and specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (ypT0/Tis ypN0). At the completion of all treatment and surgery for all enrolled participants, there will be a comparison of pCR rates between the treatment arms. pCR rates will be compared by a test of two proportions followed by logistic regression to estimate the odds ratio after adjustment for the stratification factors.
Residual cancer burden (RCB) | Up to 10 years after completion of study treatment
  Defined as a continuous measure of the extent of residual cancer after neoadjuvant chemotherapy that combines the largest diameter of the cancer in the breast, the tumor cell cellularity of the cancer, and the largest diameter and number of involved axillary lymph nodes into a single RCB score. RCB will be analyzed by comparing RCB 2-3 to RCB 0-1.
Distant relapse-free survival (DRFS) | Time from date of randomization (2nd Registration) to date of invasive distant disease recurrence or death due to any cause, assessed up to 10 years after completion of study treatment
  Analyses will be performed using log-rank testing, Cox regression, and Kaplan-Meier estimation.
Overall survival (OS) | Time from date of randomization (2nd Registration) to date of death due to any cause, assessed up to 10 years after completion of study treatment
  Analyses will be performed using log-rank testing, Cox regression, and Kaplan-Meier estimation. Will also be conducted at alpha = 0.05 (2-sided).

CONTACTS AND LOCATIONS:
Overall Officials: Erin F Cobain, Principal Investigator — SWOG Cancer Research Network
Locations (529):
- United States (527):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - City of Hope Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Huntington Memorial Hospital, Pasadena, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - City of Hope Upland, Upland, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UCI Health - Yorba Linda, Yorba Linda, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Schulze Family Foundation Cancer Clinic - Bonita Health Center, Bonita Springs, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Mease Countryside Hospital, Safety Harbor, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Ochsner LSU Health - Cancer Treatment Center, Shreveport, Louisiana
  - UM Upper Chesapeake Hematology and Oncology - Aberdeen, Aberdeen, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - The Philips Family Cancer Center, Southampton, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - UNC Health Cancer Care Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - UNC Health Cancer Care Garner, Garner, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - SWOG, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Yolanda G Barco Oncology Institute, Meadville, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Covenant Health Cancer Centers, Knoxville, Tennessee
  - Covenant Health Cancer Centers - West, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Covenant Health Oncology Group - Oak Ridge, Oak Ridge, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm